CLINICAL TRIAL: NCT00423839
Title: A Phase I Study of the Safety and Immunogenicity of MVA85A in Healthy Gambian Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AFTBVAC
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2007-01-18 (Estimated); Status verified 2006-12

CONDITIONS: Tuberculosis
Keywords: Mycobacterium tuberculosis; Antigen 85A; Modified Vaccinia Virus Ankara (MVA).
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A; Tuberculosis Vaccines

INTERVENTIONS:
Biological: MVA85A (Tuberculosis vaccine)

SUMMARY:
A Phase I study of the Safety and immunogenicity of MVA85A in healthy Gambian volunteers

DETAILED DESCRIPTION:
Study Design: The study is a non-randomized clinical trial. Twelve volunteers will be recruited. They would be given 5x107 pfu of the MVA85A vaccine intradermally. The subjects will be required to stay in the unit for an hour after the vaccination. Local and systemic adverse events would be recorded. Blood samples will be taken at the screening visit, day of immunisation, 1 week after the vaccination, then at 2, 4, 8, 12 and 24 weeks after the vaccination.

Screening:

Details of the study will be carefully discussed with the subjects and informed consent approved by the combined MRC/Gambian government ethics committee prior to any study-related evaluations being performed. The subjects that agree to enroll and have signed consent documentation will be assessed at the AFTBVAC clinic at MRC.

Entry

Subjects will be recruited at the MRC AFTBVAC clinic. Subjects will be screened in the eight weeks prior to entering the study. The screen will consist of checking subject eligibility and a full physical examination. The following will be carried out: height, weight, vital signs, haematology (haemoglobin, packed cell volume, white cell counts, platelets, blood film for malaria parasites), serum chemistry (electrolytes and creatinine, liver enzymes, serum bilirubin and proteins), Mantoux test, ELISPOT, Chest X-ray, anti-vaccinia antibodies, anti-HBV antibodies, , anti-HIV antibodies, urinalysis. All chest X-rays will be reviewed by two clinicians to confirm no radiological sign of Tuberculosis.

Evaluations during study: Scheduled follow-up:

Vaccination Day 0: after a pysician has confirmed that the volunteers are ESAT-6 and CFP-10 nagative. The following assessments will be performed pre-dosing: vital signs (20 minutes pre-dose) and blood samples collected for heamatology (haemoglobin, packed cell volume, white cell counts, platelets, blood film for malaria parasites), serum chemistry (electrolytes and creatinine, liver enzymes, serum bilirubin and proteins) and immunological assays. Provided vital signs are is satisfactory, subjects will receive the first vaccination. Subjects will have a dressing applied over the injection site, which will remain for at least one hour after the vaccination. Post vaccination vital signs will be taken at 30 and 60 minutes. Any adverse events (AEs) noted by the study personnel or described by the volunteer will be documented. Concomitant medication given will be documented. The volunteer will remain at the clinical area for one hour following vaccination and will then be allowed to return home.

Day 1 and 2: On the first and second day after vaccination subjects will be visited at home by a field worker or they will return to the clinical area. The injection site will be examined and the subjects will be questioned for AEs and use of any concomitant medications.

Day 7: Subjects will be visited at home by a field worker or they will return to the clinical area. Vital sign assessments will be performed. Blood samples will be taken for haematology(haemoglobin, packed cell volume, white cell counts, platelets, blood film for malaria parasites), serum chemistry (electrolytes and creatinine, liver enzymes, serum bilirubin and proteins) and immunological assays. The injection site will be examined and the subjects will be questioned for AEs and concomitant medications.

At day 14, 28, 56, 84 and 189, subjects will return to the clinical area. Vital sign assessments will be performed. Blood samples will be taken prior to dosing for haematology (haemoglobin, packed cell volume, white cell counts, platelets, blood film for malaria parasites), serum chemistry (electrolytes and creatinine, liver enzymes, serum bilirubin and proteins) and immunological assays. The injection site will be examined and the subjects will be questioned for AEs and concomitant medications. Day 22 and 23: On the first and second day after vaccination a field worker will visit subjects at home or they will return to the clinical area. The injection site will be examined and the subjects will be questioned for AEs and concomitant medications.

Post study Evaluations:

The injection site will be examined and the subjects asked about AEs. It is possible that they will be asked in the future to provide samples for genetic studies.

DATA COLLECTION AND MONITORING AND ADVERSE EXPERIENCE REPORTING

Records to be kept and a regulatory folder will contain:

SCC document Project Management plan Protocol with appendices Letter of ethical approval Information sheets and blank forms Signed consent forms for each subject

All filled in paper forms will be filed. Individual medical records will be filed together.

All data on the Case Report Forms (CRF) must be legibly recorded in blue or black ink or typed. A correction should be made by striking through the incorrect entry with a single line and entering the correct information adjacent to it. The correction must be initialed and dated by the investigator or a designated, qualified individual.

Any requested information that is not obtained as specified in the protocol should have an explanation noted on the CRF as to why the required information was not obtained.

Role of Data Management

The Data manager will be responsible for receiving, entering, querying, analysing, and storing the data which accrues from the study. He will be responsible for linking the epidemiological and clinical data from the field and the clinic with the laboratory data from the immunology, microbiology, haematology and genetics laboratories.

Adverse Events (AE) Reporting

Adverse events, however minor, will be recorded as observed by the Investigators or as volunteered by the subject. Full details will be documented in the CRF whether or not the Investigator or his deputies consider the event to be related to the trial substance.

Serious Adverse Events (SAE) Reporting

Serious adverse events (SAEs) that occur during the study or within six months of the final vaccination will be notified immediately (within 24 hours) by telephone to the Safety Monitor, Ethics Committee, collaborators and funding agency.

Serious adverse event are defined as an event that:

* results in death;
* is life-threatening (i.e., the subject was at risk of death at the time of the event);
* requires or prolongs in-patient hospitalization;
* results in persistent or significant disability/incapacity;
* is a congenital anomaly/birth defect;
* is a cancer.

Note:

Proven malaria events will not be included as an SAE.

Minimum details to be given in a telephone report are:

* Name of reporting doctor and contact telephone number.
* Study number.
* Nature of adverse event.
* Subject details (number, initials, sex, date of birth, weight and age).
* Date and time of event.
* Date and time of MVA85A administration and dose.
* Other drug history.
* Other relevant history.
* Outcome.
* Causality.

The event will be documented on the SAE page of the CRF and reported to the Safety Monitor, Ethics Committee, Collaborators and funding agency as appropriate. Other adverse events will be graded. After the ethics committee's response to the SAE is received, the Principal Investigator, Clinical Monitor and available co-investigators will meet to determine the future plan for the study, which could involve amending the protocol, discontinuing the vaccinations, or continuing unchanged for the other volunteers.

STATISTICAL CONSIDERATIONS

General Design Issues

A total of 12 subjects will be sufficient to provide descriptive data. As some of the subjects may drop out of the study, 12 subjects. However, only 10 individuals will be given the vaccine.

Outcomes of interest

Safety of the Vaccine

This will be determined by the degree and number of adverse events reported.

Immunogenicity of this vaccine

It is expected that the vaccine will stimulate T cell responses, which will be measured by interferon -gamma Elispot assays.

Sample Size and Accrual

Formal sample sizing calculations have not been performed but it is believed that the sample size of 10 subjects will be sufficient for this purpose.

No attempt will be made in the study to conceal the allocation group of the subjects either from the subjects themselves, the investigators or laboratory personnel.

Monitoring and Analysis

The data manager will be responsible for monitoring the trial. This will include confirming the existence of the appropriate documents in the regulatory folder and of source documents for all entered data. He would also assess the consistency of data. The data manager will be responsible for data entry and for initial analysis of the results.

The main analyses will be descriptive and comparative.

HUMAN SUBJECTS

Institutional Review Board (IRB) Review and Informed Consent

The study has been approved by the joint MRC/ Gambia government ethical committee. Written informed consent will be obtained from the subject (or parent, legal guardian, or person with power of attorney for subjects who cannot consent for themselves, such as, those below the legal age). The subject's assent must also be obtained if he or she is able to understand the nature, significance and risks associated with the study. The informed consent will describe the purpose of the study, the procedures to be followed, and the risks and benefits of participation. A signed copy of the consent form will be given to the subject (or parent or legal guardian).

Subject Confidentiality

All records will be kept in a secure place. All data on computer files will have restricted access. Clinical information will not be released without written permission of the subject, except as necessary for monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male aged 18-45 years.
* Normal medical history and physical examination. Minor physical ailments e.g. Fungal skin infections, will not be sufficient to define a physical examination as abnormal.
* Normal urine dipstick, blood count, liver enzymes, and creatinine
* Frequency <4 SFU per/well/3x105 PBMC as determined by ELISPOT with ESAT6/CFP-10 antigens and less than 100 SFU per/well/1x106 PBMC as determined by ELISPOT with PPD.
* Mantoux negative (0.0 mm induration).
* Normal Chest X-ray.
* Willing to donate blood samples as required by the protocol

Exclusion Criteria:

* Clinically significant history of skin disorder (eczema, psoriasis, etc.), allergy, immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease or neurological illness.
* Any clinical evidence of immunosuppression such as oral candida, stomatitis, aphthous or septic ulceration, septic skin lesions or any clinical or laboratory evidence of infection or immunocompromise.
* History of splenectomy
* Haematocrit of less than 30%
* Serum creatinine concentration >130mmol
* Serum ALT concentration >80IU/L
* Blood transfusion within one month of the beginning of the study
* History of vaccination with any previous experimental poxvirus vaccine
* Administration of any other vaccine or immunoglobulin within two weeks before or two weeks after vaccination.
* Positive HIV antibody test, evidence of HBV (Hepatitis B vaccination is not an exclusion criteria)..
* Current participation in another clinical trial, or within 12 weeks of this study
* Any other finding which in the opinion of the investigators would increase the risk of an adverse outcome from participation in the trial.
* Likelihood of travel away from the study area for the duration of the study
* Untreated malaria infection

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2003-03; Study Completion 2005-07

PRIMARY OUTCOMES:
Safety of the Vaccine. This will be determined by the degree and number of adverse events reported.

SECONDARY OUTCOMES:
Immunogenicity of this vaccine. It is expected that the vaccine will stimulate T cell responses, which will be measured by interferon -gamma Elispot assays.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, MD and PhD, Principal Investigator — University of Oxford
Locations (1):
- MRC Labs, Fajara, Fajara, The Gambia

REFERENCES:
- [Result] Ibanga HB, Brookes RH, Hill PC, Owiafe PK, Fletcher HA, Lienhardt C, Hill AV, Adegbola RA, McShane H. Early clinical trials with a new tuberculosis vaccine, MVA85A, in tuberculosis-endemic countries: issues in study design. Lancet Infect Dis. 2006 Aug;6(8):522-8. doi: 10.1016/S1473-3099(06)70552-7. PMID 16870530
- [Derived] Brookes RH, Hill PC, Owiafe PK, Ibanga HB, Jeffries DJ, Donkor SA, Fletcher HA, Hammond AS, Lienhardt C, Adegbola RA, McShane H, Hill AV. Safety and immunogenicity of the candidate tuberculosis vaccine MVA85A in West Africa. PLoS One. 2008 Aug 13;3(8):e2921. doi: 10.1371/journal.pone.0002921. PMID 18698342